CLINICAL TRIAL: NCT05464290
Title: Nonfat Grafting in Male and Female Genital Lichen Sclerosus
Brief Title: The Nanofat Regenerative Surgery for Management of Genital Lichen Sclerosus in Male and Female Patients
Acronym: LSNanofat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Pisa (Other); Universita di Verona (Other)
Responsible Party: Principal Investigator, Antonio Luigi Pastore, Prof, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lichen AND Nanofat grafting
Record Dates: First submitted 2022-07-05; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nanofat grafting (Experimental): The nanofat in a 10 cc syringe connected with a 23 gauge needle is used to create a lot of tunnels in the plane of the sclerotic tissues and the nanofat is delivered into the tunnels.
  Interventions: Procedure: NANOfat grafting

INTERVENTIONS:
Procedure: NANOfat grafting — The nanofat in a 10 cc syringe connected with a 23 gauge needle is then used to create a lot of tunnels in the plane of the sclerotic tissues and the nanofat is delivered into the tunnels. During injection the area is massaged to achieve complete releasing of fibrous tissue that was feel under the fingers.

SUMMARY:
Regenerative surgery is an emerging multidisciplinary field actually based on derived adipose tissue.

Autologous fat grafting was first described by Neuber in 1893 and since then it has developed over the next century. The initial goal of fat grafting was to treat volume losses created by disease or trauma. Further studies done by Zuk et al. in 2001 showed that lipoaspirate contains multipotent adipose stem cells (ADSCs) like in the bone marrow, thereby expanding opportunities in multiple fields. ADSCs have emerged as a key element of regenerative medicine surgery due to their ability to differentiate into a variety of different cell lineages. Moreover, their capacity of paracrine secretion of a broad selection of cytokines, chemokines, and growth factors make them highly clinically attractive. More specific, of particular interest are the anti-apoptotic, anti-inflammatory, proangiogenic, immunomodulatory, and anti-scarring effects that have been demonstrated for ADSCs, which effects on wound healing, soft-tissue restoration and scar remodelling.

Nanofat firstly introduced by Tonnard in 2013, is an ultra-purified adipose tissue-derived product that is devoid of mature adipocytes but rich in ADSCs and with regenerative properties.

DETAILED DESCRIPTION:
Lichen sclerosus is a chronic, inflammatory, mucocutaneous disorder of genital and extragenital skin. It was first described by Hallopeau in 1881. In 1976, the International Society for the Study of Vulvovaginal Disease concluded that the terminology LS should be adopted for men and women. Both sexes are affected, but it is 6 to 10 times more prevalent in women than in men. LS can occur at any age, but the incidence increases with age.

The aetiology of LS remains unknown thought infectious, autoimmune, and chronic irritation was investigated for the develop of LS. The autoimmune pathogenesis seems most likely. An increased incidence of autoantibodies to the extracellular matrix protein and autoantibodies to BP180 antigen in LS are reported .Other potential markers include CD4+ T-cells clones, which are found in overabundance in LS patients's tissue. and possibly promote fibroblast cell proliferation.

Risk factor to progression of LS was occlusion and exposure of urine. The susceptible epithelium may play a central role in the pathogenesis of LS. The skin may have an isotraumatopic response, to urine, feces, and other non-specific liquid irritants in occluded spaces and may play an important role in the etiology of LS in both men and women.

The Köbner phenomenon describes the occurrence of disease- specific lesions on normal appearing skin after trauma and it is described in LS. Mechanical factors like friction due to tight clothing, occlusion, surgical trauma, radiotherapy and scars are thought to play an important role in triggering and maintaining LS .

Some patients with lichen sclerosus do not have any symptoms, while most patients experience intense itching, discomfort and/or erosions/ulcers. LS is a debilitating disease, causing itch, pain, dysuria and restriction of micturition, dyspareunia, and significant sexual dysfunction in women and men. Vulvar itching, bleeding, or pain, pain during sex, skin bruising and tearing , blisters, easy bleeding from minor rubbing of the skin, trouble urinating or pain with urination, painful erections (in men). Lichen sclerosus typically has a remitting relapsing course that is complicated by permanent scarring of the affected areas.

Biopsy is worthwhile both to confirm the diagnosis and to exclude malignant change. It has been suggested that the expression of selected cellular markers (such as p53, survivin, telomerase, Ki-67, and cyclin D1) can help distinguish between indolent LS and LS with true malignant potential.

Topical and systemic treatments have been addressed but with few results. Surgery represent the solution for genital and urethral involvement. Depending on extension of genital and urethral involvement, surgical repair can range from a minimally invasive treatment to a more extensive reconstruction but still today surgery represents an open debate.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age, affected by genital lichen sclerosus

Exclusion Criteria:

* patients with age <18 y.o.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-07-25 (Estimated); Primary Completion 2022-11-20 (Estimated); Study Completion 2023-01-25 (Estimated)

PRIMARY OUTCOMES:
SURGICAL OUTCOMES | 90 days after nonfat grafting
  Visual Analog Score for pain
SURGICAL OUTCOMES | 180 days after nonfat grafting
  Visual Analog Score for pain

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Luigi Pastore, Prof, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Antonio Luigi Pastore, Latina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conde-Green A, Marano AA, Lee ES, Reisler T, Price LA, Milner SM, Granick MS. Fat Grafting and Adipose-Derived Regenerative Cells in Burn Wound Healing and Scarring: A Systematic Review of the Literature. Plast Reconstr Surg. 2016 Jan;137(1):302-312. doi: 10.1097/PRS.0000000000001918. PMID 26710034
- [Result] Doornaert M, Colle J, De Maere E, Declercq H, Blondeel P. Autologous fat grafting: Latest insights. Ann Med Surg (Lond). 2018 Oct 16;37:47-53. doi: 10.1016/j.amsu.2018.10.016. eCollection 2019 Jan. PMID 30622707